CLINICAL TRIAL: NCT05997446
Title: A Real-World Study to Observe Outcomes of Patients Undergoing Closure With the Amplatzer™ Amulet™ Left Atrial Appendage Occluder
Brief Title: Amulet™ ADVANCE LAA
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10467; CRD_1056 (Other: Abbott Medical Devices)
Record Dates: First submitted 2023-07-18; First posted 2023-08-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Left atrial appendage occlusion (LAAO) — Implantation of an Amplatzer Amulet left atrial appendage occluder

SUMMARY:
This is a prospective, multicenter, observational study intended to characterize real-world outcomes on the commercially available Amulet device in the United States. Over 600 subjects have been enrolled at 16 US clinical sites. Subjects will be followed through 24 months in accordance with each site's standard care practices.

DETAILED DESCRIPTION:
The ADVANCE LAA study is intended to characterize real-world outcomes of patients receiving the commercially available Amulet device in the United States. The Amulet device is intended to reduce the risk of thrombus embolization from the left atrial appendage (LAA) in patients who have nonvalvular atrial fibrillation (NVAF) and who are at increased risk for stroke and systemic embolism based on CHADS2 or CHA2DS2-VASc scores, are suitable for short-term anticoagulation therapy, and have appropriate rationale to seek a non-pharmacologic alternative to oral anticoagulation, taking into consideration the safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* Intended for LAAO with the Amulet device
* At least 18 years of age
* Willing and capable of providing informed consent and participating in all testing associated with this clinical study

Exclusion Criteria:

* Presence of other conditions that, in the investigator's opinion, could limit the subject's ability to participate in follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation who are at increased risk for ischemic stroke or systemic embolism.
Sampling Method: Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint: Death or complications | Within 7 days of implant or hospital discharge, whichever is later
  Composite of all-cause death, ischemic stroke, systemic embolism, or device/procedure related complications requiring an invasive surgical or percutaneous intervention within 7 days of implant or hospital discharge, whichever is later
Device closure, defined as residual jet around the device ≤ 3mm | Assessed at first trans-esophageal echocardiogram (TEE) occurring between 30-240 days post-implant.
  Device closure (defined as residual jet around the device ≤ 3mm) at the first follow-up visit documented by trans-esophageal echocardiography (TEE), as assessed by an independent core laboratory
Composite endpoint: Ischemic stroke or systemic embolism | Through 24 months
  Composite of ischemic stroke or systemic embolism through 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Cardiac Arrhythmia Research Foundation
Locations (16):
- United States (16):
  - Arizona Arrhythmia Research, Phoenix, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Baptist Medical Center, Jacksonville, Florida
  - Usman R. Siddiqui, MD, Winter Park, Florida
  - PERC - O'Fallon, O'Fallon, Illinois
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Providence Hospital, Southfield, Michigan
  - Bryan Heart, Lincoln, Nebraska
  - CHI Health Creighton University Medical Center-Bergan Mercy, Omaha, Nebraska
  - New York University Hospital, New York, New York
  - Pinnacle Health System, Mechanicsburg, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Heart Rhythm Associates, Shenandoah, Texas

IPD SHARING:
Plan to Share IPD: No